CLINICAL TRIAL: NCT00954252
Title: Placebo-Controlled, Ascending Single-Dose Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of CHF 5074 in Healthy Young Male Subjects
Brief Title: Safety, Pharmacokinetics and Pharmacodynamics Study of Treatment With CHF 5074 in Healthy Young Male Subjects
Acronym: CT01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CERESPIR (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: CCD-0814-PR-0008
Record Dates: First submitted 2009-07-31; First posted 2009-08-07 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — 1-(3',4'-dichloro-2-fluoro(1,1'-biphenyl)-4-yl)cyclopropanecarboxylic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test Article (Experimental)
  Interventions: Drug: CHF 5074
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: CHF 5074 — 1x, oral capsule, single dose
  Arms: Test Article
Drug: placebo — placebo, oral capsule, single dose
  Arms: Placebo
Drug: CHF 5074 — 2x, oral capsule, single dose
  Arms: Test Article
Drug: CHF 5074 — 4x, oral capsule, single dose
  Arms: Test Article
Drug: CHF 5074 — 8x, oral capsule, single dose
  Arms: Test Article
Drug: CHF 5074 — 16x, oral capsule, single dose
  Arms: Test Article
Drug: CHF 5074 — 24x, oral capsule, single dose
  Arms: Test Article

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of single oral doses of CHF 5074 in young healthy male volunteers.

DETAILED DESCRIPTION:
The primary endpoint of the study is to determine the maximum tolerated dose (MTD) of CHF5074 after single oral administration to young healthy male volunteers.

The secondary objective of this study is to evaluate the pharmacokinetics of CHF5074 after single oral administration to young healthy male volunteers. The secondary endpoint of this study is to verify if CHF5074 plasma levels (Cmax and AUC0-t) increase proportionally with the dose (dose-linearity).

The exploratory objective of this study is to evaluate the pharmacodynamics of CHF5074 after single oral administration to young healthy male volunteers. The respective exploratory endpoint is to assess the relationship between individual maximum CHF5074 plasma concentrations and corresponding A-beta42 plasma concentrations corrected for baseline A-beta42 levels.

ELIGIBILITY:
Inclusion Criteria:

* Subject's written informed consent is obtained prior to any study-related procedures.
* Subject is nonsmoking male between 18 and 45 years of age, inclusive.
* Subject has a body mass index between 18 and 30 kg/m2, inclusive.
* Subject is judged, by the investigator, to be in good health on the basis of medical history, complete physical examination including vital signs, 12-lead electrocardiogram (ECG) and standard laboratory tests including complete hematology, blood chemistry (glucose, creatinine, blood urea nitrogen, alanine aminotransferase, aspartate aminotransferase, albumin, alkaline phosphatase, sodium, potassium), thyroid function, urinalysis (glucose, hemoglobin, blood, proteins, pH) and fecal occult blood.
* Subject understands the procedures and agrees to participate in the study program.

Exclusion Criteria:

* Subject is mentally or legally incapacitated.
* Subject has a history of any illness that, in the opinion of the investigator and according to the protocol, might confound the results of the study or pose additional risk in administering CHF5074 to the subject.
* Subject has a medical history (within the last 10 years) of major cardiovascular, hepatic or renal disease.
* Subject has liver function test abnormalities with elevated AST or ALT greater than or equal to 2 times upper limit of normal and/or elevated bilirubin greater than or equal to 2 times upper limit of normal.
* Subject has renal function test abnormalities, including serum creatinine greater than 1.8 g/dL.
* Subject has abnormal fasting serum concentrations of TSH, T3 or T4.
* Subject has a positive result for fecal occult blood testing performed at screening.
* Subject has clinically significant abnormalities on physical examination, ECG or laboratory tests carried out at screening.
* Subject has a history of a psychiatric disorder.
* Subject has significant allergic conditions that require medical treatment or has known hypersensitivity to medications that could be activated by CHF5074 treatment.
* Subject is positive on testing for hepatitis B surface antigen, hepatitis C antibody or HIV 1 or 2 antibodies.
* Subject has donated blood within the 1 month prior to screening.
* Subject has a history of alcohol or drug abuse in the past 12 months.
* Subject used any psychoactive, recreational or prescription drug within the 4 weeks prior to study drug administration.
* Subject has used ibuprofen, sulindac sulfide, indomethacin, flurbiprofen within 2 weeks prior to study drug administration.
* Subject has used any other over-the-counter drug within 1 week prior to study drug administration Occasional treatment with acetaminophen or aspirin is permitted but must be reported to the investigator. Vitamins are permitted.
* Subject is positive on urine drug screening for drugs of abuse (cannabinoids, cocaine, opiates, amphetamines, barbiturates, benzodiazepines).
* Subject has evidence of alcohol on screening blood work and breathalyzer test.
* Subject does not agree to use a medically acceptable contraceptive (abstain from sexual intercourse, or use a condom with spermicide) for 7 days after study drug administration, or has not had a vasectomy at least 6 months prior to study participation.
* Subject is unlikely to comply with the study protocol or unable to understand the nature and scope of the study or the possible benefits or unwanted effects of the study treatments.
* Subject has participated in another investigational study within 30 days prior to screening.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2009-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Adverse Events | from Screening through Day +3

SECONDARY OUTCOMES:
Dose linearity of CHF5074 plasma levels (Cmax and AUC0-t) | Day -1 through Day +3

CONTACTS AND LOCATIONS:
Overall Officials: Joel S Ross, MD, FACP, Principal Investigator — Iberica Clinical Research Center
Locations (1):
- Iberica Clinical Research Center, Eatontown, NJ 07724, New Jersey, United States

REFERENCES:
- [Background] Lesne S, Koh MT, Kotilinek L, Kayed R, Glabe CG, Yang A, Gallagher M, Ashe KH. A specific amyloid-beta protein assembly in the brain impairs memory. Nature. 2006 Mar 16;440(7082):352-7. doi: 10.1038/nature04533. PMID 16541076
- [Background] Shankar GM, Li S, Mehta TH, Garcia-Munoz A, Shepardson NE, Smith I, Brett FM, Farrell MA, Rowan MJ, Lemere CA, Regan CM, Walsh DM, Sabatini BL, Selkoe DJ. Amyloid-beta protein dimers isolated directly from Alzheimer's brains impair synaptic plasticity and memory. Nat Med. 2008 Aug;14(8):837-42. doi: 10.1038/nm1782. Epub 2008 Jun 22. PMID 18568035
- [Background] Olson RE, Albright CF. Recent progress in the medicinal chemistry of gamma-secretase inhibitors. Curr Top Med Chem. 2008;8(1):17-33. doi: 10.2174/156802608783334088. PMID 18220929
- [Background] Lleo A. Activity of gamma-secretase on substrates other than APP. Curr Top Med Chem. 2008;8(1):9-16. doi: 10.2174/156802608783334060. PMID 18220928
- [Background] Lewis HD, Perez Revuelta BI, Nadin A, Neduvelil JG, Harrison T, Pollack SJ, Shearman MS. Catalytic site-directed gamma-secretase complex inhibitors do not discriminate pharmacologically between Notch S3 and beta-APP cleavages. Biochemistry. 2003 Jun 24;42(24):7580-6. doi: 10.1021/bi034310g. PMID 12809514
- [Background] Maillard I, Adler SH, Pear WS. Notch and the immune system. Immunity. 2003 Dec;19(6):781-91. doi: 10.1016/s1074-7613(03)00325-x. PMID 14670296
- [Background] Stanger BZ, Datar R, Murtaugh LC, Melton DA. Direct regulation of intestinal fate by Notch. Proc Natl Acad Sci U S A. 2005 Aug 30;102(35):12443-8. doi: 10.1073/pnas.0505690102. Epub 2005 Aug 17. PMID 16107537
- [Background] Searfoss GH, Jordan WH, Calligaro DO, Galbreath EJ, Schirtzinger LM, Berridge BR, Gao H, Higgins MA, May PC, Ryan TP. Adipsin, a biomarker of gastrointestinal toxicity mediated by a functional gamma-secretase inhibitor. J Biol Chem. 2003 Nov 14;278(46):46107-16. doi: 10.1074/jbc.M307757200. Epub 2003 Aug 29. PMID 12949072
- [Background] Wong GT, Manfra D, Poulet FM, Zhang Q, Josien H, Bara T, Engstrom L, Pinzon-Ortiz M, Fine JS, Lee HJ, Zhang L, Higgins GA, Parker EM. Chronic treatment with the gamma-secretase inhibitor LY-411,575 inhibits beta-amyloid peptide production and alters lymphopoiesis and intestinal cell differentiation. J Biol Chem. 2004 Mar 26;279(13):12876-82. doi: 10.1074/jbc.M311652200. Epub 2004 Jan 6. PMID 14709552
- [Background] Weggen S, Eriksen JL, Das P, Sagi SA, Wang R, Pietrzik CU, Findlay KA, Smith TE, Murphy MP, Bulter T, Kang DE, Marquez-Sterling N, Golde TE, Koo EH. A subset of NSAIDs lower amyloidogenic Abeta42 independently of cyclooxygenase activity. Nature. 2001 Nov 8;414(6860):212-6. doi: 10.1038/35102591. PMID 11700559
- [Background] Kukar T, Golde TE. Possible mechanisms of action of NSAIDs and related compounds that modulate gamma-secretase cleavage. Curr Top Med Chem. 2008;8(1):47-53. doi: 10.2174/156802608783334042. PMID 18220932
- [Background] Peretto I, La Porta E. Gamma-secretase modulation and its promise for Alzheimer's disease: a medicinal chemistry perspective. Curr Top Med Chem. 2008;8(1):38-46. doi: 10.2174/156802608783334097. PMID 18220931
- [Background] Peretto I, Radaelli S, Parini C, Zandi M, Raveglia LF, Dondio G, Fontanella L, Misiano P, Bigogno C, Rizzi A, Riccardi B, Biscaioli M, Marchetti S, Puccini P, Catinella S, Rondelli I, Cenacchi V, Bolzoni PT, Caruso P, Villetti G, Facchinetti F, Del Giudice E, Moretto N, Imbimbo BP. Synthesis and biological activity of flurbiprofen analogues as selective inhibitors of beta-amyloid(1)(-)(42) secretion. J Med Chem. 2005 Sep 8;48(18):5705-20. doi: 10.1021/jm0502541. PMID 16134939
- [Background] Imbimbo BP, Del Giudice E, Colavito D, D'Arrigo A, Dalle Carbonare M, Villetti G, Facchinetti F, Volta R, Pietrini V, Baroc MF, Serneels L, De Strooper B, Leon A. 1-(3',4'-Dichloro-2-fluoro[1,1'-biphenyl]-4-yl)-cyclopropanecarboxylic acid (CHF5074), a novel gamma-secretase modulator, reduces brain beta-amyloid pathology in a transgenic mouse model of Alzheimer's disease without causing peripheral toxicity. J Pharmacol Exp Ther. 2007 Dec;323(3):822-30. doi: 10.1124/jpet.107.129007. Epub 2007 Sep 25. PMID 17895400
- [Background] Imbimbo BP, Del Giudice E, Cenacchi V, Volta R, Villetti G, Facchinetti F, Riccardi B, Puccini P, Moretto N, Grassi F, Ottonello S, Leon A. In vitro and in vivo profiling of CHF5022 and CHF5074 Two beta-amyloid1-42 lowering agents. Pharmacol Res. 2007 Apr;55(4):318-28. doi: 10.1016/j.phrs.2006.12.010. Epub 2007 Jan 16. PMID 17292621
- [Background] Imbimbo BP, Hutter-Paier B, Villetti G, Facchinetti F, Cenacchi V, Volta R, Lanzillotta A, Pizzi M, Windisch M. CHF5074, a novel gamma-secretase modulator, attenuates brain beta-amyloid pathology and learning deficit in a mouse model of Alzheimer's disease. Br J Pharmacol. 2009 Mar;156(6):982-93. doi: 10.1111/j.1476-5381.2008.00097.x. PMID 19239474
- [Background] Sisti R, Nyska A. CHF 5074: 4-week oral toxicity study in rats followed by a 4-week recovery period. RTC Study No. 71470. February 9, 2009.
- [Background] Grassetti A, Nyska A. CHF 5074. 4 week oral toxicity study in dogs followed by a 4 week recovery period. RTC Study No. 71470. February 4, 2009.
- [Background] Cinelli S, Oberto G. CHF 5074. Unscheduled DNA Synthesis (UDS) in primary rat hepatocytes after in vivo treatment (autoradiographic methods). RTC Study No. 70270. December 4, 2008.
- [Background] Ciliutti P, Oberto G. CHF 5074. Micronucleous test in rats. RTC Study No. 70260. November 28, 2008.